CLINICAL TRIAL: NCT06184815
Title: Effectiveness of a Multidisciplinary Treatment and Structured Education for Type 1 Diabetes Patients
Brief Title: Effectiveness of a Multidisciplinary Treatment and Structured Education Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, David Sanchez Garcia, Principal investigator, Instituto Mexicano del Seguro Social
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMSST1D
Record Dates: First submitted 2023-12-15; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; Autoimmune Diseases; Diabetes; Education Programme; DSMES; Diabetes self-management education and support; T1D; Insulin-dependent diabetes; Juvenile diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Diabetes Mellitus | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The educational programme consists of 12 lessons, diabetes education slides and patient materials, with a duration of 4 months. The multidisciplinary treatment consists of 4, each one every month, consultations of specialties of nutrition, endocinrology and psychology.
Masking Description: The standard educational and treatment program consists of outpatient management and education in the office and consultation referral to nutrition and psychology with a duration of 4 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational programme 12 (Experimental): The educational programme consists of 12 lessons, diabetes education slides and patient materials, with a duration of 4 months. The multidisciplinary treatment consists of 4, each one every month, consultations of specialties of nutrition, endocinrology and psychology.
  Interventions: Behavioral: Educational programme 12
- Standard (Active Comparator): The standard educational program consists of outpatient management with diabetic education slides and material for the patient, with a duration of 4 months. Standard treatment consists of endocrinology consultation with nutrition and psychology referral if required
  Interventions: Behavioral: Standard education and treatment

INTERVENTIONS:
Behavioral: Educational programme 12 — Consists of 12 lessons, diabetes education slides and patient materials, with a duration of 4 months and multidisciplinary treatment
  Arms: Educational programme 12
Behavioral: Standard education and treatment — Outpatient management and education in the office and consultation referral to nutrition and psychology
  Other Names: Standard
  Arms: Standard

SUMMARY:
This trial compared an structured education programme and multidisciplinary treatment vs an standard treatment in type 1 diabetes patient, the Primary outcome is glycemic control at 6-month follow up and secondary outcome are cardiovascular risk factors control, diabetes related distress, anxiety and depressive symptoms, hypoglycemia awareness.

DETAILED DESCRIPTION:
Both groups will received individualized treatment in the clinic, the intervention group will consist of 12 educational sessions during 4 months, and multidisciplinary treatment each month given by endocrinology, nutrition and psychology during 4 months, the control group will received education in outpatient clinic of endocrinology and will be sent as referral to specialties of nutrition and psychology as standard follow-up of the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Diabetes duration >1 year
* BMI 18.5-40kg/m2
* A1c 6.5-13%

Exclusion Criteria:

* Pregnancy
* Dementia or severe cognitive impairment
* Uncontrolled psychiatric disorder
* Absence of >20% of the educational sessions

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Glycemic Control Measured by A1c | Baseline and 6 months
  Difference between baseline A1c and A1c at 6 month follow up

SECONDARY OUTCOMES:
Changes in Lipid Control Measured by LDLc, HDLc, non-HDLc, Triglycerides, Total Cholesterol | Baseline and 6 months
  Difference between basal lipid profile and lipid profile at 6 month follow up
Changes in insulin resistance control Measured by eGDR | Baseline and 6 months
  Difference between basal eGDR and eGDR at 6 month follow up
Changes in Mental health Measured by DDS, GAD7 and PHQ9 | Baseline and 6 months
  Difference between basal DDS, GAD7 and PHQ9 and DDS, GAD7 and PHQ9 at 6 month follow up
Changes Anthropometry Measured by BMI and WC | Baseline and 6 months
  Difference between basal BMI and WC and BMI and WC at 6 months
Changes in Glycemic Control Measured by severe hypoglycemia | Baseline and 6 months
  Difference between severe hypoglycemia in the las 6 months and severe hypoglycemia at 6 months of follow up

CONTACTS AND LOCATIONS:
Overall Officials: David Sanchez, MD, Principal Investigator — Centro Médico Nacional del Noreste Hospital de Especialidades UMAE 25 Monterrey, Mexico